CLINICAL TRIAL: NCT04999397
Title: Penetrating Cardiac Injuries: Outcome of Treatment From a Level 1 Trauma Centre in South
Status: Completed | Type: Observational
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Maeyane Stephens Moeng, Director of Trauma, University of Witwatersrand, South Africa
Other Study IDs: M180463
Record Dates: First submitted 2021-08-09; First posted 2021-08-10 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Penetrating Cardiac Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: standards clinical management — outcomes seen in cardiac injuries post clincal care

SUMMARY:
Retrospective observational study design auditing the outcomes of cardiac injuries in a single centre

DETAILED DESCRIPTION:
retrospective study over a two-year period. The demographics, injury sustained, clinical physiological parameters, mechanism of injury, injury site and patterns, outcomes and in-hospital mortality description of patients who were admitted at a single centre for further management of their cardiac injuries. Investigations performed, and procedures that were undertaken were also documented. Descriptive statistical analysis was performed. P-value of <0,05 was considered clinically significant.

ELIGIBILITY:
Inclusion Criteria: All Priority one penetrating cardiac injuries seen at CMJAH in patients who were 18 years and older -

Exclusion Criteria: Dead on arrival

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients who sustained a penetrating injury to the heart presenting at a single trauma unit
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
List injury patterns | study period (Jan 2018-Dec 2019)
  chamber involved
List of Mechanisms seen | study period (Jan 2016-Dec 2019)
  describe the type of mechanism involved in injury
outcomes | study period (Jan 2016-Dec 2019)
  overall inhospitable mortality and outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Maeyane Moeng, Principal Investigator — University of Witwatersrand, South Africa
Locations (1):
- Charlotte Maxeke Johanneburg Academic Hospital, Johannesburg, Gautheng, South Africa

IPD SHARING:
Plan to Share IPD: No